CLINICAL TRIAL: NCT06982287
Title: A Retrospective Real-World Study on the Efficacy and Safety of Anlotinib Hydrochloride Combined With Immunotherapy as Maintenance Therapy Following First-Line Chemoimmunotherapy in Treatment-Naïve Patients With Extensive-Stage Small Cell Lung Cancer (ES-SCLC) (ALTER-L059)
Brief Title: A Retrospective Real-World Study on the Efficacy and Safety of Anlotinib Hydrochloride Combined With Immunotherapy Maintenance Therapy Following Standard Chemoimmunotherapy for ES-SCLC (ALTER-L059)
Status: Not yet recruiting | Type: Observational
Sponsor: Yong Fang (Other)
Responsible Party: Sponsor-Investigator, Yong Fang, professor, Sir Run Run Shaw Hospital
Organization: Sir Run Run Shaw Hospital (Other)
Other Study IDs: ALTER-L059
Record Dates: First submitted 2025-05-06; First posted 2025-05-21 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Small Cell Lung Cancer Extensive Stage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental Group: patients treated with anlotinib Hydrochloride combined with immunotherapy maintenance therapy following standard chemoimmunotherapy.

SUMMARY:
This retrospective real-world study aims to evaluate the efficacy and safety of anlotinib hydrochloride combined with immunotherapy as maintenance therapy following standard chemoimmunotherapy in extensive-stage small cell lung cancer (ES-SCLC).The study population consists of treatment-naïve ES-SCLC patients who did not progress after induction chemoimmunotherapy and subsequently received maintenance therapy with anlotinib plus immunotherapy. The primary objectives are progression-free survival (PFS)，overall survival (OS)

, and safety.

DETAILED DESCRIPTION:
This multicenter study seeks to retrospectively analyze medical records (January 2022-December 2024) of extensive-stage small cell lung cancer (ES-SCLC) patients treated with anlotinib hydrochloride (12/10/8 mg doses) alongside immune maintenance therapy after first-line chemoimmunotherapy in real-world clinical settings. Key data points will encompass demographics, baseline disease characteristics, treatment regimens, efficacy outcomes (e.g., objective response rate, progression-free survival), and adverse event profiles. Eligible patients must have received anlotinib for ≥6 weeks and possess evaluable radiographic assessments. The primary objectives are to assess the clinical effectiveness and safety of this combination strategy in ES-SCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 years or older;
2. Histologically or cytologically confirmed extensive-stage small cell lung cancer (ES-SCLC) (per the Veterans Administration Lung Study Group [VALG] staging criteria);
3. Patients who previously received chemotherapy for limited-stage SCLC must have undergone curative-intent therapy (e.g., chemotherapy, radiotherapy, or chemoradiotherapy) and have a treatment-free interval of at least 6 months from the end of prior therapy (last chemotherapy cycle or radiotherapy) to the diagnosis of ES-SCLC;
4. At least one measurable target lesion (per RECIST version 1.1 criteria);
5. No disease progression after receiving 4-6 cycles of first-line chemoimmunotherapy induction therapy for ES-SCLC;
6. ECOG performance status: 0-2;
7. Life expectancy ≥3 months.

Exclusion Criteria:

1. Patients with limited-stage SCLC who previously received chemotherapy and underwent curative-intent therapy (e.g., chemotherapy, radiotherapy, or chemoradiotherapy) but experienced disease recurrence within 6 months after completion of prior therapy;
2. Patients with limited-stage SCLC who previously received immunotherapy agents (e.g., PD-1/PD-L1 inhibitors) or anti-angiogenic agents (e.g., Anlotinib, Apatinib, Bevacizumab);
3. Patients with extensive-stage small cell lung cancer (ES-SCLC) who developed disease progression during induction therapy with a standard chemoimmunotherapy regimen;
4. Active autoimmune diseases requiring systemic therapy (e.g., disease-modifying agents, corticosteroids, or immunosuppressants) within 2 years prior to the first dose;
5. Patients with coagulation dysfunction, defined as an International Normalized Ratio (INR) >1.5 or activated partial thromboplastin time (APTT) >1.5 × upper limit of normal (ULN), and/or those with a bleeding tendency;
6. Patients deemed by the inves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with treatment-naïve extensive-stage small cell lung cancer (ES-SCLC) who achieved non-progression after chemoimmunotherapy induction and received anlotinib plus immunotherapy maintenance therapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS2 | up to 12 months
  Progression-free survival from the initiation of anlotinib combined with immunotherapy maintenance treatment.

SECONDARY OUTCOMES:
PFS | up to 12 months
  Progress free survival
6-month PFS rate | up to 12 months
  Progress free survival rate at 6 months after diagnosis.
12-month PFS rate | up to 12 months
  Progress free survival rate at 12 months after diagnosis.
OS | From diagnosis until death (up to 24 months)
  Overall Survival
6-month OS rate | up to 12 months
  Overall survival rate at 6 months after diagnosis.
12-month OS rate | up to 24 months
  Overall survival rate at 12 months after diagnosis.
Incidence of Treatment-Emergent Adverse Events | up to 24 months
  Record Adverse Events (AEs) according to CTCAE (V5.0). Record and analyze the number of abnormal data.

IPD SHARING:
Plan to Share IPD: No